CLINICAL TRIAL: NCT02280954
Title: A Pilot and Feasibility Study of Intraoperative Imagery of Solid Tumors With Indocyanine Green
Brief Title: Indocyanine Green for Solid Tumors
Acronym: 818012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sunil Singhall, Assistant Proffesor of Medicine, Assistant Proffesor of Surgery, Director Thoracic Surgery Research Lab, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 818012; 818012 [UPenn IRB Protocol#] (Other: IRB)
Record Dates: First submitted 2013-11-21; First posted 2014-11-03 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Solid Tumor; Neoplasms
Keywords: Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG injection group (Experimental): This group will receive a single dose of ICG, infused over 40 minutes. During surgery, they will be imaged with a camera and an imaging probe the investigators have developed.
  Interventions: Drug: Indocyanine Green (ICG)

INTERVENTIONS:
Drug: Indocyanine Green (ICG)
  Other Names: ICG

SUMMARY:
According to the World Health Organization, cancer is a leading cause of death in men and women, accounting for 7.6 million deaths (around 13% of all deaths) in 2008. Surgery remains the best option for patients presenting with operable Stage I or II cancers, however the five year survival rate for these candidates remains at a dismally low. The high rates of recurrence suggest that surgeons are unable to completely detect and remove primary tumor nodules in a satisfactory manner as well as lingering metastases in sentinel lymph nodes. By ensuring a negative margin through near-infrared imagery it would be possible for us to improve the rates of recurrence from patients and thus overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Patients presenting with a solid tumor presumed to be resectable cancer and are at risk for local recurrence on pre-operative assessment
3. Good operative candidate as determined by the treating physician and multidisciplinary team
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

1. Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery
2. Subjects with a history of iodide allergies
3. Vulnerable patient populations

   1. People who would be easily lost to follow up
   2. Patients unable to participate in the consent process (children and neonates).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The ability of the imaging system to detect the expression of the ICG in the nodule/mass (i.e tumor) and discern the uptake of the dye by the tumor. | Before surgery

SECONDARY OUTCOMES:
The number of participants that will have an adverse reaction to the ICG. | Day 1-Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Predina JD, Newton AD, Corbett C, Xia L, Shin M, Sulfyok LF, Okusanya OT, Cengel KA, Haas A, Litzky L, Kucharczuk JC, Singhal S. A Clinical Trial of TumorGlow to Identify Residual Disease During Pleurectomy and Decortication. Ann Thorac Surg. 2019 Jan;107(1):224-232. doi: 10.1016/j.athoracsur.2018.06.015. Epub 2018 Jul 17. PMID 30028985
- [Derived] Lee JYK, Pierce JT, Thawani JP, Zeh R, Nie S, Martinez-Lage M, Singhal S. Near-infrared fluorescent image-guided surgery for intracranial meningioma. J Neurosurg. 2018 Feb;128(2):380-390. doi: 10.3171/2016.10.JNS161636. Epub 2017 Apr 7. PMID 28387632